CLINICAL TRIAL: NCT00409734
Title: Frequency of Formula Change Prior to the Accurate Diagnosis of Pyloric Stenosis
Status: Completed | Type: Observational
Sponsor: Maimonides Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 06/09/VA03
Record Dates: First submitted 2006-12-08; First posted 2006-12-11 (Estimated); Last update posted 2018-08-17 (Actual); Status verified 2018-08

CONDITIONS: Pyloric Stenosis
Keywords: pyloric; stenosis
MeSH Terms: conditions — Pyloric Stenosis; Constriction, Pathologic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- Children with pyloric stenosis: Male or female children age two to nine weeks with history of vomiting and feeding intolerance, and abdominal sonogram showing presence of pyloric stenosis
  Interventions: Behavioral: Children with pyloric stenosis
- Children without pyloric stenosis: Male or female children age two to nine weeks without pyloric stenosis admitted to the hospital for other reasons
  Interventions: Behavioral: Children without pyloric stenosis

INTERVENTIONS:
Behavioral: Children with pyloric stenosis — Both cohorts' feeding habits will be observed and recorded for the purposes of comparison
  Groups: Children with pyloric stenosis
Behavioral: Children without pyloric stenosis — Both cohorts' feeding habits will be observed and recorded for the purposes of comparison
  Groups: Children without pyloric stenosis

SUMMARY:
The purpose of this study is to determine if there is an increase in the frequency of formula change in patients with pyloric sctenosis prior to being correctly diagnosed.

DETAILED DESCRIPTION:
The study can be described as a prospective and retrospective study in which information will be gathered from questionnaires, analysis of medical records, and the information obtained from diagnostic procedures (i.e. Laboratory results, ultrasonography). The time of enrollment will be at the time of hospital admission for the study group and the control group. The length of time for which the patient will be involved with the study will coincide with the length of stay in the hospital. This will be a single center trial involving Maimonides Medical center. Approximately 50-100 subjects will be enrolled overall to give the study more credibility.

Methods and Procedures:

1. Study Participants: All patients admitted to Maimonides Medical Center with a diagnosis of pyloric stenosis two to nine weeks of age. Patients will be excluded from the study if there is a diagnosed milk allergy, history of prior abdominal surgery, or history of prematurity or metabolic disease. Controls will be made up of the same age range, with similar exclusion criteria, and will consist of patients admitted for other reasons than listed above, such as bronchiolitis and rule out sepsis.

2: Data: Data will be received through the completion of questionnaire.

3. Data collection and processing: Questionnaire responses will be analyzed and the responses will be statistically analyzed for correlation.

Benefits: Through participation in this study, patients may help future patients diagnosed with pyloric stenosis be brought to the attention of a medical professional.

Risks: With maintenance of confidentiality, risks to participants in this study are negligible.

ELIGIBILITY:
Inclusion Criteria:

* infants ages 2-9 weeks

Exclusion Criteria:

* infant not ages 2-9 weeks or patients with history of medical problems

Ages: 2 Weeks to 9 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Male and female children age 2 weeks to 9 weeks, either with pyloric stenosis or without
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2006-09-28 (Actual); Primary Completion 2008-12-08 (Actual); Study Completion 2008-12-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Beth Loveridge-Lenza, DO, Principal Investigator — Maimonides Medical Center; Maya Greenberg, DO, Principal Investigator — Maimonides Medical Center
Locations (1):
- Maimonides Medical Center, Brooklyn, New York, United States